CLINICAL TRIAL: NCT02443025
Title: Teens Against Tobacco Use: A Model for Universal Tobacco Prevention and Youth Advocacy
Acronym: TATU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Paso del Norte Health Foundation (Other)
Responsible Party: Principal Investigator, Louis D. Brown, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-14-0729
Record Dates: First submitted 2015-05-01; First posted 2015-05-13 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Tobacco Smoking Behavior
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Classes receive anti-tobacco presentations from Teens Against Tobacco Use members
  Interventions: Behavioral: Teens Against Tobacco Use
- Wait list control (No Intervention): Classes continue as usual without receiving anti-tobacco presentations from Teens Against Tobacco Use members until the end of the year, when data collection is complete.

INTERVENTIONS:
Behavioral: Teens Against Tobacco Use — Teens Against Tobacco Use teen teachers develop and then deliver anti-tobacco presentations to the target population of younger students.
  Arms: Intervention

SUMMARY:
This study evaluates the efficacy of Teens Against Tobacco Use anti-tobacco presentations on tobacco use susceptibility in 4th-8th grade. Classrooms are randomly assigned to either receive a series of two presentations or wait listed to receive them later in the school year.

DETAILED DESCRIPTION:
The investigators will collaborate with Austin High School, Wiggs Middle School, and Guillen Middle School of the El Paso Independent School District to implement smoke free youth coalitions as an after school activity. The coalitions will follow the Teens Against Tobacco Use (TATU) model developed by the American Lung Association, the American Cancer Society, and the American Heart Association. Participating youth will be trained to develop and deliver anti-tobacco presentations to younger students. Each school will have a separate youth coalition operating under the guidance of an adult coordinator. High school youth will present to middle school classes, whereas middle school youth will present to 4th and 5th graders.

To evaluate the efficacy of the smoke-free presentations, the investigators will first match pairs of classrooms willing to have a presentation and then randomly assign one classroom in each pair to either receive the presentation first (intervention condition) or later in the school year (control condition). Following a presentation to a classroom in the intervention condition, investigators will administer a brief survey about tobacco to students in both the intervention class and its matched control class, who have not yet received a presentation. Analyses will compare intervention and control classrooms on smoking susceptibility, perceptions of harm from tobacco use, tobacco industry perceptions, and social norms on tobacco use.

ELIGIBILITY:
Inclusion Criteria:

* 4th to 8th grade student
* Classroom must be willing to be randomly assigned to either receive presentations earlier in the school year or late in the school year

Exclusion Criteria:

* Classes in participating schools that are not in the 4th to 8th grade
* Students not able to read English or Spanish

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2414 (Actual)
Dates: Start 2014-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Standardized Tobacco Susceptibility as assessed by 12 likert scale items drawn primarily from the global youth tobacco survey | within 24 hours of receiving presentation
  Tobacco susceptibility captures the likelihood of using tobacco in the future. It is a continuous variable that will be standardized, so outcomes will represent standard deviation unit differences in tobacco susceptibility.

CONTACTS AND LOCATIONS:
Overall Officials: Louis D Brown, Ph.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, School of Public Health, El Paso Regional Campus, El Paso, Texas, United States

REFERENCES:
- [Derived] Brown LD, Bandiera FC, Harrell MB. Cluster Randomized Trial of Teens Against Tobacco Use: Youth Empowerment for Tobacco Control in El Paso, Texas. Am J Prev Med. 2019 Nov;57(5):592-600. doi: 10.1016/j.amepre.2019.06.013. Epub 2019 Sep 26. PMID 31564599